CLINICAL TRIAL: NCT02413983
Title: Comparison of Postoperative Outcome of Hepatectomy for Living Donors According to Three Different Incision: Conventional Incision vs Minimal Incision vs Transverse Incision Assisted by Laparoscopy
Brief Title: Comparison of Postoperative Outcome of Hepatectomy for Living Donors According to Three Different Incision
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gaab Soo Kim, Samsung Medical Center, Samsung Medical Center
Other Study IDs: 2015-01-016-002
Record Dates: First submitted 2015-04-02; First posted 2015-04-10 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Healthy Donors for Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CI (conventional incision): The living liver donors underwent hepatectomy using right subcostal incision with a midline extension (conventional incision)
  Interventions: Procedure: hepatectomy conventional incision
- MI (midline incision): The living liver donors underwent hepatectomy using upper midline incision (10cm) without laparoscopic assistance
  Interventions: Procedure: hepatectomy midline incision
- TI (transverse incision): The living liver donors underwent hepatectomy using transverse incision with laparosocpic assistance
  Interventions: Procedure: hepatectomy transverse incision

INTERVENTIONS:
Procedure: hepatectomy conventional incision — This study was a single center, nonrandomized, observational comparative analysis of 3 different surgical technique. Three surgical teams operated alternately at our center, and donors undergoing hepatectomy via three different incision
  Groups: CI (conventional incision)
Procedure: hepatectomy midline incision
  Groups: MI (midline incision)
Procedure: hepatectomy transverse incision
  Groups: TI (transverse incision)

SUMMARY:
Living donor liver transplantation (LDLT) is an important option for patients with end-stage liver disease requiring liver transplantation. When performing LDLT, the safety and well being of donors is of the utmost importance. The conventional incision for donor hepatectomy is a right subcostal incision with a midline extension up to xiphoid. Minimally invasive liver surgery throughout a single 10 cm upper midline incision without laparoscopic assistance has been widely applied and considered to be safe and effective. Recently, laparoscopic and minimally invasive living donor hepatectomy via transverse incision has been suggested to reduce morbidity and the invasiveness of living donor hepatectomy. Although minimally invasive approach has become the surgical method of choice for many transplant centers, little data on comparing the impact of all three different type incision in living liver donors. In our center, the investigators have adopted three different incision according to surgical teams. The investigators undertook this study with the aims of comparing the pain and quality of life of donors according to type of three different incisions and assessing any benefits to the donor due to the smaller midline incision during the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status I-II,
* adult undergoing hepatectomy for living donors

Exclusion Criteria:

* known allergy to any of the drugs used in this study,
* bleeding diathesis,
* neurologic dysfunction (preexisting lower limb neurological deficit),
* recent systemic or local infections,
* history of drug use, or
* under treatment with opioids because of chronic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was a single center, non-randomized, observational comparative analysis of 3 different surgical technique. The living liver donors underwent hepatectomy using three different type of incisions; 1) right subcostal incision with a midline extension 2) upper midline incision without laparoscopic assistance 3) transverse incision with laparosocpic assistance
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
donor recovery/quality of life (as measure bye the quality of recovery [OoR] score) | postoperative 7 day
  QoR (quality of recovery) -15, has recently been developed, which can provide an extensive yet efficient evaluation of postoperative recovery from the patient's perspective [8]. The QoR-15 is an abbreviation of the longer and more comprehensive QoR-40 [15], and includes questions on pain, physical comfort, physical independence, psychological support and emotional state, and can be completed in approximately 2 minutes.

SECONDARY OUTCOMES:
consumption of analgesics on postoperative day | 1, 4, 8, 24, 48 and 72 h after surgery
discomfort related to the scar | postoperative 7 day
  abdominal wall sensorineural deficits (numbness and differences in tactile and temperature sensations) and tightness around the scar
discomfort related to the scar | postoperative 30 day
  abdominal wall sensorineural deficits (numbness and differences in tactile and temperature sensations) and tightness around the scar
side effects (nausea, vomiting, back pain, pruritus) | 1, 4, 8, 24, 48 and 72 h after surgery
  nausea, vomiting, back pain, pruritus
donor recovery/quality of life (as measure bye the quality of recovery [OoR] score) | postoperative 30 day
  QoR (quality of recovery) -15, has recently been developed, which can provide an extensive yet efficient evaluation of postoperative recovery from the patient's perspective [8]. The QoR-15 is an abbreviation of the longer and more comprehensive QoR-40 [15], and includes questions on pain, physical comfort, physical independence, psychological support and emotional state, and can be completed in approximately 2 minutes.
assessment of subjective pain (as measured by numeric rating scale [NRS]) on postoperative day | 1, 4, 8, 24, 48 and 72 h after surgery
  numeric rating scale (NRS) in which; 0 = no pain and 100 = worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea